CLINICAL TRIAL: NCT01385670
Title: InterSEPT: In-Tunnel SeptRx European PFO Trial: A Prospective, Multi-Center Study to Evaluate the Safety and Performance of the SeptRx IPO PFO Closure System
Brief Title: InterSEPT: In-Tunnel SeptRx European PFO Trial
Acronym: InterSEPT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SeptRx, Inc. (Industry)
Responsible Party: Beverly Tang, SeptRx, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InterSEPT
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Foramen Ovale, Patent; Heart Defects, Congenital; Heart Septal Defects
Keywords: Patent Foramen Ovale; PFO
MeSH Terms: conditions — Foramen Ovale, Patent; Heart Defects, Congenital; Heart Septal Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Transcatheter PFO closure with the SeptRx Intrapocket PFO Occluder (IPO) — Transcatheter PFO closure

SUMMARY:
The objective of this study is to determine the safety, performance, and effectiveness of the SeptRx IPO PFO Closure System in the treatment of Patent Foramen Ovale (PFO) in patients who are amenable to percutaneous closure of their PFO defects.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥ 18 years of age and ≤ 70 years of age
* The patient is willing to comply with specified follow-up evaluations
* The patient or legally authorized representative has been informed of the nature of the study, agrees to its provisions and has been provided written Notice of Informed Consent, approved by the appropriate Ethics Committee (EC)
* PFO flat width of 4-14mm (approximate PFO balloon diameter of 2.5-9mm) and PFO length of 4-20mm

Exclusion Criteria:

* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure
* Other medical illness (e.g., cancer, known malignancy, congestive heart failure, organ transplant recipient or candidate) or known history of substance abuse (alcohol, cocaine, heroin etc.)
* Known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, Nitinol, and/or contrast sensitivity that cannot be adequately pre-medicated
* Currently participating in another investigational study, or participation in another clinical trial in the previous 3 months
* PFO flat width <4mm or >14mm to begin the trial. PFO flat width <4mm or >19mm when the second size device is ready
* PFO length <4mm or >20mm
* Active endocarditis, active bacterial infection, or other infection producing bacteremia or sepsis
* History of chronic or sustained arrhythmia
* Congenital or structural heart disease other than PFO
* Thrombus at the intended site of implant or documented venous thrombosis in venous access
* Severe pulmonary hypertension
* Vascular anatomy unable to accommodate the appropriate-sized sheath for device introduction
* Acute appendicitis
* Confinement to bed (increased risk for clot formation)
* Prior cardiac surgery, including implantation of active cardiac devices

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Safety: Major Adverse Events defined as composite rate of all death, stroke, device embolization, tamponade, and device related re-intervention or surgery | One (1) month

SECONDARY OUTCOMES:
Efficacy: Device success defined as PFO closure at 6 months post procedure by transesophageal echocardiography (TEE) with contrast valsalva bubble study. | Six (6) months

CONTACTS AND LOCATIONS:
Locations (2):
- ICPS: Institut Jacques Cartier, Massy, France
- CardioVasculäres Centrum Frankfurt, Frankfurt, Germany

REFERENCES:
- [Background] Zimmermann WJ, Heinisch C, Majunke N, Staubach S, Russell S, Wunderlich N, Sievert H. Patent foramen ovale closure with the SeptRx device initial experience with the first "In-Tunnel" device. JACC Cardiovasc Interv. 2010 Sep;3(9):963-7. doi: 10.1016/j.jcin.2010.04.019. PMID 20850097